CLINICAL TRIAL: NCT02967809
Title: Usefulness of an Ultraportative Ultrasound Device in the Management of Intra Hospital Emergencies
Status: Completed | Type: Observational
Sponsor: Hospital Nord (Other)
Responsible Party: Sponsor
Other Study IDs: 00010254 --- 2016 --- 122
Record Dates: First submitted 2016-11-14; First posted 2016-11-18 (Estimated); Last update posted 2020-04-27 (Actual); Status verified 2020-04

CONDITIONS: Respiratory Failure; Failure; Cardiac
MeSH Terms: conditions — Respiratory Insufficiency; Heart Failure | interventions — Ultrasonography

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Month
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- final diagnosis after portable echography: Experimental group: final diagnosis after portable cardiac echograph examination
  Interventions: Device: echography
- final diagnosis without portable echography: Group control: Final diagnosis for patient ( same medical condition and history) hospitalized in units without portable cardiac echograph examination avaible

INTERVENTIONS:
Device: echography — cardiac and pulmonary echography
  Groups: final diagnosis after portable echography

SUMMARY:
Estimate if the use of a portable cardiac echograph for intra-hospital Emergencie improves the performances diagnose in the bed of patient in department of conventional medicine.

The concordance between the initial medical diagnosis (previous the utilsation of portable echograph) and the final diagnosis (after portable echograph utisation) will be evaluated. These evaluation will be performed after retrospective review of the medical files

ELIGIBILITY:
Inclusion Criteria:

* respiratory or cardiac distress

Exclusion Criteria:

* pulmonary or cardiac patient transplant morphologic abnormalities Patient in rescucitation care unit

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient suffering of respiratory or cardiac distress
Sampling Method: Non-Probability Sample
Enrollment: 172 (Actual)
Dates: Start 2016-10 (Actual); Primary Completion 2018-11 (Actual); Study Completion 2019-09 (Actual)

PRIMARY OUTCOMES:
Concordance between initial medecial diagnosis and final diagnosis | 1 day
  Concordance between the initial medical diagnosis at the bedside in ward and the definitive diagnosis after retrospective review of the medical files between two groups : one with an ultraportative echograph (POCUS group) and a control (without ultraportative group). The percentage of adequate initiale diagnosis at the bedside.

CONTACTS AND LOCATIONS:
Overall Officials: Marc Leone, MD, Principal Investigator — DAR Nord
Locations (1):
- Departement anesthesie reanimation hopital nord, Marseille, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Zieleskiewicz L, Lopez A, Hraiech S, Baumstarck K, Pastene B, Di Bisceglie M, Coiffard B, Duclos G, Boussuges A, Bobbia X, Einav S, Papazian L, Leone M. Bedside POCUS during ward emergencies is associated with improved diagnosis and outcome: an observational, prospective, controlled study. Crit Care. 2021 Jan 22;25(1):34. doi: 10.1186/s13054-021-03466-z. PMID 33482873